CLINICAL TRIAL: NCT05521815
Title: Effect of Early Coma Arousal Therapy on Conscious Level Recovery and Cognition in Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mustafa Samir Mohamed Amin Sayed, Senior Physiotherapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 54531
Record Dates: First submitted 2022-08-23; First posted 2022-08-30 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Traumatic Brain Injury With Loss of Consciousness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): The group that are going to receive the coma arousal therapy program
  Interventions: Other: Coma arousal therapy
- Control group (Placebo Comparator): This group will receive only traditional treatment program
  Interventions: Other: Selected physiotherapy program

INTERVENTIONS:
Other: Coma arousal therapy — early coma arousal therapy program in addition to selected physical therapy program (positioning, breathing exercise, passive movement of the four limbs).
  Arms: Study group
Other: Selected physiotherapy program — selected physiotherapy program only (positioning, breathing exercise, passive movement of the four limbs).
  Arms: Control group

SUMMARY:
PURPOSE:

The aim of this study is to investigate the effect of early coma arousal therapy on conscious level and cognitive function in sever traumatic brain injury patients.

BACKGROUND:

Traumatic brain injury (TBI) could be simply defined as an alteration in brain function due to external forces and is considered as one of the leading cause of death and disability worldwide, especially among young adults and the elderly. Current estimates imply that annual incidence of TBI is 50-60 million worldwide, and specifically for Europe and USA, 0.5% of Europeans and 1.1% of Americans are experiencing a TBI each year.

The original scale has since been revised and is known as the Rancho Los Amigos Revised Scale (RLAS-R). One of the limitations of the original eight level scale was that it did not accurately reflect the individuals with higher levels of recovery. Two more levels were added to the initial eight level Ranchos Scale to create a more comprehensive ten level scale named the Rancho Los Amigos Revised Scale (RLAS-R).

DETAILED DESCRIPTION:
The aim of this study is to examine the early effect of coma arousal therapy on Conscious Level Recovery and Cognition in Traumatic Brain Injury. forty two patients will be selected and they will be assigned in to two different group, a study group where will they recieve coma arousal therapy in addition to conventional therapy and a control group where they will recieve only the conventional physical therapy program.

ELIGIBILITY:
Inclusion criteria:

1. Both genders.
2. Traumatic brain injury with GCS score 3-12.
3. Age range from 20-50 years old.
4. Must be medically stable post trauma 29

Exclusion Criteria:

1. Patient with other neurological deficits or orthopedic abnormalities that causing disability.
2. Patients with pre injury psychiatric disorders.
3. Patients with pre injury cognitive disorders.
4. Patients who performed surgery post traumatic brain injury.
5. Patients not taking the same medications.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
conscious level | One and half year
  is defined as the state of awareness of the self and environment with appropriate arousal or wakefulness. conscious level will be measured using glascow coma scale (GCS), which is a scale used to objectively describe the extent of impaired consciousness in all types of acute medical and trauma patients. The highest possible GCS score is 15, and the lowest is 3. A score of 15 means you're fully awake, responsive and have no problems with thinking ability or memory. Generally, having a score of 8 or fewer means you're in a coma. The lower the score, the deeper the coma is.
Cognition | One and half year
  'cognition' refers to all the processes by which the sensory input is transformed, reduced, elaborated, stored, recovered, and used. It is concerned with these processes even when they operate in the absence of relevant stimulation, as in images and hallucinations. cognition will be measured using Rancho Los Amigos Revised Scale (RLAS-R), its a scale used by both medical and rehabilitation providers to measure and track cognitive recovery after traumatic brain injury. It is a 10-point scale where Level I indicates No response/total assistance and Level X indicates Purposeful, appropriate/ modified independent.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr el Aini hospital, Cairo, Egypt